CLINICAL TRIAL: NCT02757846
Title: Quantitative Imaging for Evaluation of Response to Cancer Therapies
Brief Title: Radiomics of Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: Eastern Hepatobiliary Surgery Hospital (Other); Guangdong Provincial People's Hospital (Other); Henan Provincial People's Hospital (Other); West China Hospital (Other); Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Chongwei Chi, Ph.D, Quantitative Imaging for Evaluation of Response to Cancer Therapies, Chinese Academy of Sciences
Other Study IDs: 20160427ABCD
Record Dates: First submitted 2016-04-28; First posted 2016-05-02 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: Radiomics; prognosis; medical images; Hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
We propose a radiomics approach to identify prognostic biomarkers of HCC and provide patients with some reasonable advice for their therapies.

DETAILED DESCRIPTION:
Radiomics is emerging fields that is based on quantitative analysis of medical images. Tri-phasic CT images are currently the standard imaging modality for the management of HCC. Our goal is to improve treatment decisions of HCC patients through better understanding of their prognosis based on radiomics modeling of HCC. Radiomics is defined as the extraction of quantitative image features from medical images. We will use triphasic CT data of at least 200 patients and develop a robust strategy to extract imaging features from CT. We will use deep learning in the form of a Convolutional Neural Network to segment HCC lesions and use image feature extraction algorithms with supervised classification to predict prognosis.

ELIGIBILITY:
Inclusion Criteria:

* The purpuse of our research is to improve treatment ,therefore we have no creteria.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Currently, a cohort of 20 patients has already been collected from the collaborating hospitals. Next, the 5 hospitals will collect at least 1200 patients within 1-2 years and up to 6000 patients during the full course of the project (5 years).
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2017-04; Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
quantitative image features extracted from CT images can be used as imaging marker for prognosis | five(year)

CONTACTS AND LOCATIONS:
Overall Officials: di dong, PhD, Study Director — Chinese Academy of Sciences
Locations (1):
- Key Laboratory of Molecular Imaging, Chinese Academy of Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shen W, Zhou M, Yang F, Yang C, Tian J. Multi-scale Convolutional Neural Networks for Lung Nodule Classification. Inf Process Med Imaging. 2015;24:588-99. doi: 10.1007/978-3-319-19992-4_46. PMID 26221705
- [Background] Wilkerson MD, Hayes DN. ConsensusClusterPlus: a class discovery tool with confidence assessments and item tracking. Bioinformatics. 2010 Jun 15;26(12):1572-3. doi: 10.1093/bioinformatics/btq170. Epub 2010 Apr 28. PMID 20427518
- [Background] Sanson M, Marie Y, Paris S, Idbaih A, Laffaire J, Ducray F, El Hallani S, Boisselier B, Mokhtari K, Hoang-Xuan K, Delattre JY. Isocitrate dehydrogenase 1 codon 132 mutation is an important prognostic biomarker in gliomas. J Clin Oncol. 2009 Sep 1;27(25):4150-4. doi: 10.1200/JCO.2009.21.9832. Epub 2009 Jul 27. PMID 19636000
- [Background] Cui Y, Jia J. Update on epidemiology of hepatitis B and C in China. J Gastroenterol Hepatol. 2013 Aug;28 Suppl 1:7-10. doi: 10.1111/jgh.12220. PMID 23855289
- [Background] Zhu F, Shi Z, Qin C, Tao L, Liu X, Xu F, Zhang L, Song Y, Liu X, Zhang J, Han B, Zhang P, Chen Y. Therapeutic target database update 2012: a resource for facilitating target-oriented drug discovery. Nucleic Acids Res. 2012 Jan;40(Database issue):D1128-36. doi: 10.1093/nar/gkr797. Epub 2011 Sep 24. PMID 21948793
- See also: A Website from Key Laboratory of Molecular Imaging, Chinese Academy of Sciences — http://www.mitk.net/